CLINICAL TRIAL: NCT02097693
Title: Effect of Deep Brain Stimulation in the Globus Pallidus Internus on Quality of Life in Young Patients With Dyston-dyskinetic Cerebral Palsy
Brief Title: Effect of DBS on Quality of Life in Dyskinetic Cerebral Palsy
Acronym: STIM-CP
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: University Hopsital Schleswig Holstein Campus Lübeck (Other); Boston Scientific Corporation (Industry); University Hsopital of Magdeburg (Unknown); University Hospital of Munich (Unknown); Schoen Klinik Vogtareuth (Unknown); University Hospital of Tübingen (Unknown); Heinrich-Heine University, Duesseldorf (Other); Hannover Medical School (Other); University Hospital of Kiel (Unknown); University Hospital of Würzburg (Unknown); University Hospital of Freiburg (Unknown); University Hospital Berlin Charite (Unknown)
Responsible Party: Principal Investigator, Anne Koy, Priv.-Doz. Dr. med. Anne Koy, University of Cologne
Other Study IDs: Uni-Koeln-1603
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dyskinetic Cerebral Palsy Due to Perinatal Hypoxia
Keywords: DBS; quality of life; dystonia; dyskinetic cerebral palsy
MeSH Terms: conditions — Dystonia; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA-plasma for DYT1-testing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- dyston-dyskinetic cerebral palsy: Young patients with dyston-dyskinetic cerebral palsy who receive DBS in the GPi

SUMMARY:
There are limited therapeutical options for patients with secondary dystonia due to cerebral palsy. Pharmacotherapy is often without effect, or side effects are severe. Meanwhile deep brain stimulation (DBS) has proven to be a safe and effective therapy for patients with parkinson´s disease or primary / idiopathic dystonia. Experiences with DBS in patients with dyskinetic cerebral palsy are limited with heterogeneous data.

With STIM-CP we investigate the effect of DBS on quality of life in young patients with a dyskinetic movement disorder (dyskinetic cerebral palsy) due to perinatal hypoxic brain injury. Additionally, the effect of DBS on motor development, speech, memory, attention, cognition and pain perception will be assessed.

DETAILED DESCRIPTION:
In total, 20 patients aged 7-18 years diagnosed with dyskinetic cerebral palsy due to perinatal asphyxia, who will receive DBS, should be included. 11 German DBS-centres will participate in the trial. Effects of DBS will be assessed up to 36 months after Initial Implantation.

There are two preoperative visits (screening and baseline) and nine postoperative visits (implantation, 3-, 6-, 9-, 12-, 24- and 36-moths follow-up). We assume that DBS reduces the severity of dystonia and improves the quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* The treating physician has chosen GPi-DBS for the treatment of the secondary dystonia caused by cere-bral palsy in this patient
* Patient and/or legal representative, if the patient is underaged or not capable to give consent himself, have chosen GPi-DBS as treatment
* The consent to participate in the trial of the underaged patient, if he is capable to understand the study requirements, is required
* Age at enrolment 7-18 years
* Diagnosis of secondary dystonia due to cerebral palsy caused by perinatal hypoxic injury
* Anti-dystonic pharmacotherapy insufficient (e.g. Jankovic J. Medical treatment of dystonia. Movement disorders, Vol. 28, No. 7, 2013) 67
* Stable anti-dystonic medication over the last 30 days
* Globus pallidus internus (pars posterior) and thalamus (motor part) intact on MRI (not older than 2 years - if possible)
* No fixed severe skeletal deformations with loss of function, which need immediate orthopaedic surgical intervention
* Sufficient compliance of the patient or the legal representative if the patient is underaged or not capable to give consent himself to take part in the study
* Informed consent to take part in the study from patient and/or legal representative if the patient is underaged or not capable to give consent himself
* Patient and/or legal representative if the patient is underaged or not capable to give consent himself, understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* • Patients with known primary (e.g. DYT1) or idiopathic dystonia

  * Severe axial hypotonia with total loss of head control (e.g. absence of control at "upper thoracic level" in the SATCo score) (medication effect excluded)
  * Fixed hemi-dystonia
  * Severe spasticity in knee- and elbow-flexors and -extensors (Modified Ashworth Scale >3)
  * Fixed severe skeletal contractions with loss of function which require immediate orthopaedic surgical intervention
  * Patients with other severe concurrent neurological disease (e. g. brain tumor, neurodegenerative diseases, trauma etc.)
  * Condition likely to require use of MRI in the future
  * Any intracranial abnormality or medical condition that would contraindicate DBS surgery
  * Any findings in neuropsychological screening assessments that would contraindicate DBS surgery
  * Any current drug and / or alcohol abuse
  * Any history of frequent grand-mal seizures without response to anticonvulsive treatment
  * Any other active implanted device (e.g. Cochlear implant, pacemaker), whether turned on or off, would be allowed provided that they do not interfere with functioning of the device.
  * Any previous brain surgery that would interfere with the placement of the leads or the functioning of the device.
  * A history of neurostimulation intolerance in any area of the body.
  * Currently on any anticoagulant medications that cannot be discontinued during perioperative period.
  * Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.
  * Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days; any other trial participation should be approved by the Principal Investigator.
  * A female that is breastfeeding or of child bearing potential with a positive urine pregnancy test or - if a person is sexually active - not using sufficient contraception with a Pearl Index of less than 1% including all forms of hormonal contraception ("antibaby-pill", hormonal plaster, NuvaRing®, Implanon®, hormonal depot injections, contraceptive coil), the tubal ligature (female sterilization). Alternatively, the female of child bearing potential is sexually abstinent.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | CPCHILD 12 months after DBS
  Difference in CPCHILD before and 36 months on DBS (response=improvement > 10%)

SECONDARY OUTCOMES:
Burke-Fahn-Marsden-Dystonia Rating Scale movement and disability | 0, 6, 12, 24 and 36 months after DBS
  Assessment of the severity of dystonia
Dyskinesia Impairment Scale | 0, 12, 24 and 36 months
  Assessment of the severity of chorea and dystonia
Tardieu Scale | 0 and 12 months after DBS
  Assessment of the severity of spasticity
Frenchay Dysarthria Assessment | 0, 12, 24 and 36 months after DBS
  Assessment of speech and swallowing
SF-36 | 0, 6, 12, 24 and 36 months after DBS
  Assessment of Quality of life
Strengths and Difficulties Questionnaire | 0, 6, 12, 24 and 36 months after DBS
  Assessment of mood and attention
Snijders-Oomen-Non-Verbal-Intelligence Test (SON-R) | 0 and 12 months
  Assessment of Cognition
Attentional Network Test (ANT) | 0 and 12 months after DBS
  Assessment of Attention
Non-Verbal-Learning Test (NVLT) | 0 and 12 months after DBS
  Assessment of cognition
Wong Baker Faces | 0, 6, 12, 24 and 36 months after DBS
  Assessment of pain
Family Scale (FaBel) | 0, 6, 12, 24 and 36 months after DBS
  Assessment of the burden for caregivers
Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | 0, 6, 24 and 36 months after DBS
  Assessment of quality of life
Canadian Occupational Performance Measure (COPM) | COPM 0 and 12 months after DBS
  Assessment of activities of daily living
Gross Motor Function Measure (GMFM-66) | GMFM-66 0 and 12 months after DBS
  Assessment of physical disability
Gross Motor Function Classification System (GMFCS) | GMFCS 0, 12, 24 and 36 months after DBS
  Degree of physical impairment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Koy, MD, Principal Investigator — University Hospital Cologne, Germany
Locations (1):
- University Hospital Cologne, Cologne, Northern Westfalia, Germany

REFERENCES:
- [Derived] Koy A, Kuhn AA, Huebl J, Schneider GH, van Riesen AK, Eckenweiler M, Rensing-Zimmermann C, Coenen VA, Krauss JK, Saryyeva A, Hartmann H, Haeussler M, Volkmann J, Matthies C, Horn A, Schnitzler A, Vesper J, Gharabaghi A, Weiss D, Bevot A, Marks W, Pomykal A, Monbaliu E, Borck G, Mueller J, Prinz-Langenohl R, Dembek T, Visser-Vandewalle V, Wirths J, Schiller P, Hellmich M, Timmermann L; STIM-CP investigators. Quality of Life After Deep Brain Stimulation of Pediatric Patients with Dyskinetic Cerebral Palsy: A Prospective, Single-Arm, Multicenter Study with a Subsequent Randomized Double-Blind Crossover (STIM-CP). Mov Disord. 2022 Apr;37(4):799-811. doi: 10.1002/mds.28898. Epub 2021 Dec 29. PMID 34967053